CLINICAL TRIAL: NCT04695678
Title: Epidemiological Multicohort Study of Latent COVID-19 Infections in Residents and Staff of Nursing Homes in the City of Solingen
Brief Title: Epidemiological Multicohort Study of Latent COVID-19 Infections
Status: Completed | Type: Observational
Sponsor: Wissenschaftliches Institut Bethanien e.V (Other)
Responsible Party: Sponsor
Other Study IDs: WI-2020179
Record Dates: First submitted 2020-12-11; First posted 2021-01-05 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- residents and staff of all nursing homes in Solingen: each study participant receives a single nasal/pharyngeal swab
  Interventions: Diagnostic Test: COVID-19 nasal/pharyngeal swab
- staff of one single nursing home in Solingen: each study participant receives a weekly nasal/pharyngeal swab for six months
  Interventions: Diagnostic Test: COVID-19 nasal/pharyngeal swab

INTERVENTIONS:
Diagnostic Test: COVID-19 nasal/pharyngeal swab — each study participant receives a nasal/pharyngeal swab

SUMMARY:
Cross-sectional study to detect latent COVID-19 infections in residents and staff of old people's and nursing homes in the city of Solingen with a prospective follow-up of 6 months in a subgroup.

DETAILED DESCRIPTION:
Particular interest is being paid to old people's and nursing homes during the COVID-19 pandemic, as people at particular risk are to be found there. Therefore, the health department of the city of Solingen will carry out extensive testing of both staff and residents for COVID-19 in this sensitive area. The scientific institute Bethanien für Pneumologie e.V. would like to collect and evaluate the data and test results collected in the process in order to record the occurrence of infections in this area and to obtain information on possible routes of infection and the effectiveness of hygiene measures taken. The aims of the study are:

1. Prevalence of latent COVID-19 infections at one point in time among residents and staff of old people's and nursing homes in Solingen.
2. Prevalence of latent COVID-19 infections over a period of 6 months among staff of a single nursing home (=subgroup)
3. Analysis of transmission pathways of the virus in a nursing home
4. Analysis of the effectiveness of hygiene measures taken
5. Analysis of risk factors (previous illnesses, medication, etc.)

ELIGIBILITY:
Inclusion Criteria:

* informed consent of the test person or the legally authorised guardian

Exclusion Criteria:

* missing consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All residents and staff in the nursing homes in Solingen who consent to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1462 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of latent COVID-19 infections at one point in time among residents and staff of all old people's and nursing homes in Solingen. | baseline
  number of positive COVID-19 tests
Prevalence of latent COVID-19 infections over a follow-up period of 6 months among staff of one single nursing home | 6 months
  number of positive COVID-19 tests

SECONDARY OUTCOMES:
Analysis of risk factors (previous illnesses, medication...) | 6 months
  analysis of risk factors for a COVID-19 infection

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Randerath, Principal Investigator — Krankenhaus Bethanien Solingen
Locations (1):
- Institut für Pneumologie an der Universität zu Köln / Wissenschaftliches Institut Bethanien für Pneumologie e.V., Solingen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No